CLINICAL TRIAL: NCT01650051
Title: A Double-Blind, Randomized, Multi-Center, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Phenazopyridine Hydrochloride Tablets, USP 200 mg as an Analgesic for Short-Term Treatment in Female Subjects Suffering From Moderate-to-Severe Pain and Burning Upon Urination Associated With Uncomplicated Urinary Tract Infections (uUTI)
Brief Title: Safety and Efficacy of Phenazopyridine Hydrochloride Tablets, USP 200 mg as an Analgesic for Short-Term Treatment in Female Subjects Suffering From Moderate-to-Severe Pain and Burning Upon Urination Associated With Uncomplicated Urinary Tract Infections (uUTI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-PHN-004
Record Dates: First submitted 2012-07-19; First posted 2012-07-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Uncomplicated Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo of Phenazopyridine Hydrochloride Tables, USP 200 mg (Placebo Comparator)
  Interventions: Drug: Placebo of Phenazopyridine Hydrochloride Tables, USP 200 mg
- Phenazopyridine Hydrochloride Tables, USP 200 mg (Experimental)
  Interventions: Drug: Phenazopyridine Hydrochloride Tables, USP 200 mg

INTERVENTIONS:
Drug: Placebo of Phenazopyridine Hydrochloride Tables, USP 200 mg — Deep brown maroon colored, film coated round biconvex tablet debossed 'AN" obve '2' on one side and plain on the other side.
  Arms: Placebo of Phenazopyridine Hydrochloride Tables, USP 200 mg
Drug: Phenazopyridine Hydrochloride Tables, USP 200 mg — Deep brown maroon colored, film coated round biconvex tablet debossed 'AN" obve '2' on one side and plain on the other side.
  Arms: Phenazopyridine Hydrochloride Tables, USP 200 mg

SUMMARY:
The primary objective is to evaluate the safety and efficacy of Phenazopyridine HCl Tablets, USP 200 mg as a short term analgesic treatment of pain upon urination associated with Uncomplicated Urinary Tract Infections (uUTI).

The secondary exploratory objective is to evaluate safety and efficacy of Phenazopyridine HCl Tablets, USP 200 mg as a short term analgesic treatment of burning upon urination associated with uUTI.

DETAILED DESCRIPTION:
Subjects will make separate self-assessments for severity of pain and burning upon urination using the NRS and self-assessments of their discomfort using the GSAS at designated intervals for 24 hours. Subjects will rate the effectiveness of the study medication using the SASMS at a designated interval for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide and understand written informed consent for the study.
* Is a female 18 years of age or older.
* Has a clinical diagnosis of uncomplicated urinary tract infection (uUTI).
* Has a reported history indicating a diagnosis of cystitis or urethritis.
* Has a positive urine dipstick test showing the presence of nitrate or leukocyte esterase.
* Has moderate to severe pain (score of 4 to 10 inclusive on the NRS) and burning (score of 4-10, inclusive on the NRS) upon urination.
* Is willing and able to understand and comply with the requirements of the study.
* Each female subject of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years) must have a negative urine pregnancy test at Screening and must be willing to use an acceptable form of birth control during the study. For the purpose of this trial, the following are considered acceptable methods of birth control: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (eg, condom and spermicide), contraceptive injection (Depo-provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control should the subject become sexually active.

Exclusion Criteria:

* Is pregnant or breastfeeding during the study.
* Has a diagnosis of a urinary tract or kidney disorder that is not a uUTI. Has a diagnosis of pyelonephritis (kidney infections when lower uUTI spreads to the upper tract).
* Has taken an analgesic within 1 day prior to Visit 1.
* Has taken any systemic anti-infectives within 7 days prior to Visit 1.
* Has a history of G-6-PD deficiency or hemolytic anemia.
* Has a known history of anatomical genitourinary (GU) anomalies or GU surgery within 6 months prior to Visit 1.
* Has a chronic infection of the urinary tract requiring an intravenous pyelogram (IVP), ultrasound, or cystoscopy.
* Is unable to comprehend the language of the informed consent and the self-evaluation scales.
* Has serious acute illness (e.g., pneumonia) or an untreated or unstable medical illness that would likely interfere with assessments of uUTI.
* Has received an investigational medication as part of a drug trial within 3 months prior to Visit 1.
* Is currently participating in any other clinical study.
* Has a history of severe drug allergy or hypersensitivity, including to phenazopyridine HCl or to any component of the study medications.
* Consumes excessive amounts of alcohol, abuses drugs, or has any condition that would compromise compliance with this protocol.
* Previous participation in this study.
* Any clinically significant condition or situation, that in the opinion of the Investigator would interfere with the study evaluations or optimal participation in the study.
* Prior use of phenazopyridine product within 3 years of enrollment.
* Is an employee or direct relative of the study site or Investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Self-assessments | Designated Intervals for 24 hours
  The difference between baseline NRS for pain at 0 hours and the NRS for pain score at each scheduled time will be calculated to obtain Pain Intensity Difference (PID) at each time point 92, 4, 6, 8, 16 and 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Symbio, LLC, Port Jefferson, New York, United States